CLINICAL TRIAL: NCT05423106
Title: A Phase 1, Blinded, Randomized, Placebo-controlled, First-in-human Study of Orally Administered JNJ-64457744 to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics After Single and Multiple Ascending Doses
Brief Title: A Single and Multiple Ascending Dose Study of JNJ-64457744
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic business decision, not due to safety concerns
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CR109208; 64457744HPB1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-06-06; First posted 2022-06-21 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; tenofovir alafenamide; entecavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1: JNJ-64457744 or Placebo (Single Ascending Dose [SAD] Cohorts A-F) (Experimental): Non-Asian healthy participants will receive a SAD of either JNJ-64457744 or matching placebo as an oral formulation under fasted conditions on Day 1. Cohort F will be optional.
  Interventions: Drug: JNJ-64457744; Drug: Placebo
- Part 1: JNJ-64457744 (Cohorts G-H) (Experimental): Non-Asian healthy participants will receive 3 single doses of JNJ-64457744 as an oral formulation in 3 intervention periods (to assess inter-subject PK-PD) matching the doses evaluated in Cohorts A, C and E for Cohort G and Cohorts B, D and F for Cohort H, under fasted conditions on Day 1. Cohort H will be optional for Intervention period 3.
  Interventions: Drug: JNJ-64457744
- Part 1: JNJ-64457744 or Placebo (Cohort I) (Experimental): Non-Asian healthy participants who previously received study intervention under fasted conditions will receive either JNJ-64457744 or matching placebo as an oral formulation (depending upon what was administered previously in Cohorts A to F) under fed conditions on Day 1.
  Interventions: Drug: JNJ-64457744; Drug: Placebo
- Part 1: JNJ-64457744 or Placebo (Cohort J) (Experimental): Asian healthy participants will receive a single dose at one single dose level of either JNJ-64457744 or matching placebo, as an oral formulation, under fasted conditions on Day 1.
  Interventions: Drug: JNJ-64457744; Drug: Placebo
- Part 1: JNJ-64457744 (Cohort K) (Experimental): Optional Cohort K: Non-Asian healthy participants will receive an oral formulation of JNJ-64457744 in the first intervention period and will cross over to receive the other formulation during the second intervention period, under fasted conditions on Day 1.
  Interventions: Drug: JNJ-64457744
- Part 2 JNJ-64457744 or Placebo (Experimental): Chronic hepatitis B participants who are virologically suppressed on nucleos(t)ide analog (NA) treatment (tenofovir disoproxil fumarate [TDF], tenofovir alafenamide [TAF] and entecavir [ETV]) will receive a single dose at one single dose level of either JNJ-64457744 or matching placebo as an oral formulation, under fasted condition on Day 1.
  Interventions: Drug: JNJ-64457744; Drug: Placebo; Drug: Tenofovir Disoproxil Fumarate (TDF); Drug: Tenofovir Alafenamide (TAF); Drug: Entecavir (ETV)
- Part 3: JNJ-64457744 or Placebo (Multiple Ascending Doses [MADs]) (Experimental): Participants will receive MADs of either JNJ-64457744 or matching placebo once weekly under fasted conditions as an oral formulation.
  Interventions: Drug: JNJ-64457744; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64457744 — JNJ-64457744 will be administered as oral solution.
  Arms: Part 1: JNJ-64457744 (Cohorts G-H); Part 1: JNJ-64457744 or Placebo (Cohort I); Part 1: JNJ-64457744 or Placebo (Cohort J); Part 1: JNJ-64457744 or Placebo (Single Ascending Dose [SAD] Cohorts A-F); Part 2 JNJ-64457744 or Placebo; Part 3: JNJ-64457744 or Placebo (Multiple Ascending Doses [MADs])
Drug: Placebo — Placebo will be administered as an oral formulation.
  Arms: Part 1: JNJ-64457744 or Placebo (Cohort I); Part 1: JNJ-64457744 or Placebo (Cohort J); Part 1: JNJ-64457744 or Placebo (Single Ascending Dose [SAD] Cohorts A-F); Part 2 JNJ-64457744 or Placebo; Part 3: JNJ-64457744 or Placebo (Multiple Ascending Doses [MADs])
Drug: Tenofovir Disoproxil Fumarate (TDF) — TDF tablet will be administered orally
  Arms: Part 2 JNJ-64457744 or Placebo
Drug: Tenofovir Alafenamide (TAF) — TAF tablet will be administered orally.
  Arms: Part 2 JNJ-64457744 or Placebo
Drug: Entecavir (ETV) — ETV tablet will be administered orally.
  Arms: Part 2 JNJ-64457744 or Placebo
Drug: JNJ-64457744 — JNJ-64457744 will be administered as oral tablet.
  Arms: Part 1: JNJ-64457744 (Cohort K)

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of: single ascending dose (SAD) and multiple ascending dose (MAD) administration of JNJ-64457744, administered to healthy adult participants (Part 1 and Part 3), including a cohort of Asian participants (Part 1); and after single dose administration of JNJ-64457744 to chronic hepatitis B (CHB) participants who are virologically suppressed on nucleos(t)ide analog (NA) treatment (tenofovir disoproxil fumarate [TDF], tenofovir alafenamide [TAF], or entecavir [ETV]) (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Normal left ventricular heart function as defined as left ventricular ejection fraction (LVEF) greater than or equal to (>=) 5 percent (%), as assessed by 2 dimension electrocardiogram (2DECHO) at screening
* All women must have a negative urine pregnancy test at screening and Day -1 (of each intervention period, if applicable)
* A woman must not be of childbearing potential
* Part 1 and 3: Must have an estimated creatinine clearance greater than (>) 80 milliliter (mL) per minute at screening, calculated by the modification of diet in renal disease (MDRD) formula
* Part 2: Must have chronic HBV infection. HBV infection must be documented by serum HBsAg positivity at screening
* Must be fully vaccinated against coronavirus disease 2019 (COVID-19) at least 2 weeks prior to screening calculated by the modification of diet in renal disease (MDRD) formula
* Participants in Cohorts A-I and K in Part 1 must not have maternal and paternal parents and/or grandparents of Asian ethnicity (that is, China, Japan, Korea as confirmed by interview) Participants in Cohort J must have maternal and paternal parents and grandparents of Asian ethnicity (that is, China, Japan, Korea as confirmed by interview)

Exclusion Criteria:

* History of cardiac arrhythmias (example, extrasystole, tachycardia at rest), history of risk factors for Torsades de Pointes syndrome (example, hypokalemia, family history of long QT syndrome) or history or other clinical evidence of significant or unstable cardiac disease (example, angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia, coronary heart disease, and/or clinically significant electrocardiogram ([ECG] abnormalities), moderate to severe valvular disease or uncontrolled hypertension at screening. Any evidence of second and third degree heart block or right bundle branch block is also exclusionary
* Participants with abnormal sinus rhythm (heart rate less than [<] 45 or > 100 beats per minute [bpm]), QT corrected for heart rate according to Fridericia's formula (QTcF) > 450 milliseconds (ms) for male participants and > 470 ms for female participants, QRS >= 120 ms, PR interval >220 ms, abnormal conduction, or any other clinically significant abnormalities on a 12-lead ECG at screening
* Family history of inherited mitochondrial disorders such as inherited mitochondrial myopathy, mitochondrial encephalomyopathy with lactic acidosis and stroke-like episodes (MELAS) syndrome
* Known allergies, hypersensitivity, or intolerance to JNJ-64457744 or its excipients
* History of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Part 1, 2 and 3: Number of Participants With Serious Adverse Events (SAEs) | Up to Week 8
  SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; suspected transmission of any infectious agent via medicinal product; or any important medical events.
Part 1, 2 and 3: Number of Participants With SAEs by Severity | Up to Week 8
  SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; suspected transmission of any infectious agent via medicinal product; or any important medical events. Severity will be graded according to the Division of Division of Acquired Immunodeficiency Syndrome (DAIDS) grading table where Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Potentially Life-threatening.
Part 1, 2 and 3: Number of Participants With Clinical Laboratory Abnormalities | Up to 8 weeks
  Number of participants with clinical laboratory abnormalities (including hematology, biochemistry, coagulation, urinalysis) will be reported.
Part 1, 2 and 3: Number of Participants With Clinical Laboratory Abnormalities by Severity | Up to 8 weeks
  Number of participants with clinical laboratory abnormalities (including hematology, biochemistry, coagulation, urinalysis) will be reported. Severity will be graded according to the Division of AIDS (DAIDS) grading table where Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Potentially Life-threatening.
Part 1, 2 and 3: Number of Participants With Electrocardiograms (ECGs), Echocardiography, Vital Signs and Physical Examination Abnormalities | Up to Week 8
  Number of participants with abnormalities in ECGs, echocardiography, vital signs and physical examination will be reported.
Part 1, 2 and 3: Number of Participants With Electrocardiograms (ECGs), Echocardiography, Vital Signs and Physical Examination Abnormalities by Severity | Up to 8 weeks
  Number of participants with abnormalities in ECGs, echocardiography, vital signs and physical examination will be reported. Severity will be graded according to the Division of AIDS (DAIDS) grading table where Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Potentially Life-threatening.
Part 1, 2 and 3: Plasma concentration of JNJ-64457744 | Up to Week 8
  Plasma concentration of JNJ-64457744 will be reported.

SECONDARY OUTCOMES:
Part 1: Plasma Concentration of JNJ-64457744: Within-Participant Analysis | Up to 5 weeks
  Plasma concentration of JNJ-64457744 assessed within-participant after administration of 3 different single doses under fasted conditions will be reported.
Part 1: Plasma Concentration of JNJ-64457744 Under Fed and Fasted Condition | Up to 5 weeks
  Plasma Concentration of JNJ-64457744 under fed and fasted conditions will be reported.
Part 1: Plasma Concentration of JNJ-64457744 Under Fasted Condition in Healthy Adult Asian Participants | Up to 5 weeks
  Plasma concentration of JNJ-64457744 under fasted conditions in healthy adult Asian participants will be reported.
Part 1: Plasma Concentration of JNJ-64457744 Formulation Under Fasted Conditions | Up to 5 weeks
  Plasma Concentration of JNJ-64457744 formulation as compared with an oral solution formulation under fasted conditions will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (1):
- New Zealand Clinical Research, Grafton, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency